CLINICAL TRIAL: NCT05522660
Title: A Multicentre Randomised Open-label Phase III Study of Stereotactic Radiosurgery, in Addition to Standard Systemic Therapy for Patients With Metastatic Melanoma or Newly Diagnosed Metastatic NSCLC and Asymptomatic or Oligo-symptomatic Brain Metastases
Brief Title: Immunotherapy or Targeted Therapy With or Without Stereotactic Radiosurgery for Patients With Brain Metastases From Melanoma or Non-small Cell Lung Cancer
Acronym: USZ-STRIKE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: USZ Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 19-21
Record Dates: First submitted 2022-08-23; First posted 2022-08-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer; Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — Radiosurgery; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard systemic treatment with stereotactic radiosurgery (SRS) (Experimental): Arm A
  Interventions: Radiation: Stereotactic radiosurgery; Drug: Immune checkpoint inhibitor
- Standard systemic treatment without stereotactic radiosurgery (Active Comparator): Arm B
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Radiation: Stereotactic radiosurgery — Depending on the investigator's preference, the following standard of care fractionation schedules are recommended: 1x 18-22 Gy, 3x 9 Gy or 5x 6 Gy. Fractionated stereotactic radiotherapy is favoured in principle, but not mandated, for postoperative radiotherapy and for metastases with a diameter of >20 mm or for >4 brain metastases.
  For patients randomised to Arm A, radiotherapy should be initiated within 14 days after randomisation.
  Arms: Standard systemic treatment with stereotactic radiosurgery (SRS)
Drug: Immune checkpoint inhibitor — Systemic therapy follows the current standard of care, according to the type of the primary tumour.
  * For patients with melanoma, with or without BRAF-mutation, systemic therapy consists of
    * an approved immune-checkpoint inhibition combination therapy (cohort 1a) or
    * an approved immune-checkpoint inhibition monotherapy (cohort 1b).
  * For patients with NSCLC and a targetable oncogenic driver alteration (cohort 2a), systemic therapy consists of an approved targeted therapy (for example: EGFR-, ALK- or ROS1-targeted treatment).
  * For patients with NSCLC without a targetable oncogenic driver alteration (cohort 2b), systemic therapy consists of an approved immune-checkpoint inhibition therapy (with or without chemotherapy).
  Other Names: standard of care treatment

SUMMARY:
The primary objective of the study is to assess the efficacy in terms of CNS-specific PFS of the combination of standard systemic treatment plus SRS vs. standard systemic treatment alone in patients with newly diagnosed and untreated (except for surgery) asymptomatic or oligosymptomatic brain metastases from melanoma or NSCLC. This proposed randomised phase III clinical study addresses one of the most controversial issues in the current approach to patients with brain mets: the timing of SRS in patients eligible for systemic immune checkpoint inhibition or targeted therapy in order to guide therapeutic options as to what strategy allows the best compromise between best survival and best QoL.

ELIGIBILITY:
Most important inclusion criteria:

* Newly diagnosed, previously untreated (except for surgery, see below) asymptomatic or oligo-symptomatic brain metastases, e.g., controlled symptomatic seizure disorder. Note: patients with neurological symptoms or signs that require more than a stable dose of 4 mg dexamethasone equivalent for more than one week are not considered oligo-symptomatic.
* Requirements for brain metastases:
* Brain metastases must be previously untreated, except for surgery.
* Prior surgery (including biopsies, resection, and cyst aspiration) for brain metastases is allowed. Residual and measurable disease after surgery is not required, but surgery must have confirmed the diagnosis. An MRI performed within 72 hours post-surgery should be available.
* Number and size of metastases at diagnosis of brain metastases:

  * Maximum 1-10 brain metastases at screening
  * At least one brain metastasis must be of ≥5 mm in diameter
  * In case of 1-4 brain metastases:
  * Longest diameter of largest brain metastasis must be ≤30 mm
  * In case of 5-10 brain metastases:
  * Largest metastasis must be ≤10 mL in volume and longest diameter must be ≤30 mm
  * Maximum cumulative brain metastases volume must be ≤30 mL
* Primary disease of histologically confirmed (from primary tumour or from a metastatic lesion, including in the brain) melanoma or NSCLC
* Requirements for patients with melanoma:
* Prior treatment, including treatment with immune-checkpoint inhibitors is permitted, but brain metastases must be newly diagnosed and previously untreated (except for surgery).
* BRAF-mutation status, locally assessed, should be known (previous adjuvant BRAF-targeted therapy is allowed).
* Requirements for patients with NSCLC:
* Newly diagnosed, treatment-naïve (except for prior surgery) metastatic NSCLC, with or without a targetable oncogenic driver alteration.
* Known PD-L1 expression status (from primary tumour or from a metastatic lesion, including brain)
* Known driver mutation status (from primary tumour or from a metastatic lesion, including brain).
* Age of 18 years or older
* Karnofsky performance status of 60 or more
* Life expectancy >12 weeks
* Patients must be candidates for systemic treatment, within the defined cohorts (melanoma: cohorts 1a and 1b; NSCLC: cohorts 2a and 2b).
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 7 days before randomisation.
* Written IC for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention.

Most important exclusion criteria:

* Confirmed or probable leptomeningeal metastases according to EANO ESMO criteria
* Symptomatic brain metastases at time of randomisation, e.g., neurological symptoms or signs that require more than a stable dose of 4 mg dexamethasone equivalent for more than one week.
* Patients must be off steroids or on a stable dose of ≤4 mg dexamethasone equivalent at randomisation.
* Patients experiencing seizures controlled by anti-epileptic drugs are eligible.
* Prior whole brain irradiation or focal radiation therapy to the brain
* Prior systemic treatment for brain metastases
* Contra-indication for SRS
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CNS-specific PFS, locally assessed as per iRANO criteria | from date of randomization until the date of documented CNS-specific progression, assessed up to 42 months
  The primary objective of the study is to assess the efficacy in terms of CNS-specific progression-free survival (PFS) of the combination of standard systemic treatment plus SRS versus standard systemic treatment alone in patients with newly diagnosed and untreated (except surgery) asymptomatic or oligo-symptomatic brain metastases from melanoma or non-small cell lung cancer, with indication for systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, MD, Study Chair — University of Zurich; Rolf Stahel, MD, Study Chair — ETOP IBCSG Partners Foundation
Locations (15):
- Italy (6):
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Instituto Oncologico Veneto IRCCS, Padua
  - Santa Maria della Misericordia Hospital, Perugia
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - Policlinico Umberto 1, Rome
  - Azienda ospedaliero-universitaria Senese Siena, Siena
- NKI-AVL, Amsterdam, Netherlands
- Spain (3):
  - Vall Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital La Fe, Valencia
- Switzerland (3):
  - Inselspital, Bern
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich, Zurich
- United Kingdom (2):
  - Royal Marsden (Sutton), London
  - Christie NHS Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No